CLINICAL TRIAL: NCT03525067
Title: Colonization of Bile Ducts and Postoperative Infectious Complications of Pancreaticoduodenectomies
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2016/PERTEK/ELR
Record Dates: First submitted 2018-04-26; First posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Pancreatic Cancer; Sepsis; Bile Duct Cancer; Duodenal Cancer; Bile Duct; Obliteration; Post-Op Complication; Post-Op Infection; Fistula, Biliary; Fistula; Delayed Gastric Emptying
MeSH Terms: conditions — Pancreatic Neoplasms; Sepsis; Bile Duct Neoplasms; Duodenal Neoplasms; Postoperative Complications; Biliary Fistula; Fistula; Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Bile Samples: Patients underwent pancreaticoduodenectomy who had intraoperative bile sampling for bacterial examination.
  Interventions: Other: Bile sampling for bacterial examination

INTERVENTIONS:
Other: Bile sampling for bacterial examination — At the beginning of pancreaticoduodenectomy, patients had bile sampling from the gallbladder or from the common bile duct for bacterial examination and study of susceptibility to antibiotics.

SUMMARY:
The aim of the present prospective study was, first, to verify the correlation between biliary colonization and postoperative infectious complications, and secondarily to asses morbidity and mortality for patients who underwent pancreaticoduodenectomy.

The hypothesis is that a proportion of post-operative infections after pancreaticoduodenectomy is due to bacteria that colonize the bile ducts during the preoperative period.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy is part of the curative treatment of periampullary neoplasms. Postoperative mortality for this procedure is between 1 and 5 %, and morbidity ranging from 30 to 50%. Infectious complications, with pancreatic fistula and gastric delayed empting, are an important part of this morbidity, affecting nearly 35% of patients.

One of the risk factors of infectious complications is the presence of a preoperative obstructive jaundice, due to obstruction of bile ducts by the tumor. In this case, it is proposed to perform a preoperative drainage of the bile ducts, preferably by endoscopic procedure (ERCP), associated with the placement of a endoprosthesis. However, this procedure is controversial, this one increasing postoperative morbidity, and in particular the rate of infectious complications. One explanation of these events is the bacteriological contamination of the bile ducts during the endoscopic procedure. In addition, it has been observed for the patients who have benefited from preoperative drainage, the biliary flora is predominantly polymicrobial and may contain multiresistant nosocomial germs, unlike patients who have not benefited from this procedure, whose biliary flora is predominantly sterile or monomicrobial. This colonization by multiresistant germs may have consequences in the postoperative period, in fact, up to 49% of the germs found in the bile samples are also found in the samples taken during postoperative infectious events. This microbial release could make it more difficult to take care of postoperative infections, with less efficacy of conventional antibiotic treatments.

The aim of the present prospective study was, first, to verify the correlation between biliary colonization and postoperative infectious complications, and secondarily to asses morbidity and mortality in patients who underwent pancreaticoduodenectomy. Patients whit colonized bile and patients with sterile bile were compared for these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18
* patients underwent programmed pancreaticoduodenectomy

Exclusion Criteria:

* Patients underwent emergency pancreaticoduodenectomy (delay less than 48 hours)
* Patients had not been taken of a biliary sample in intraoperative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18, patients underwent programmed pancreaticoduodenectomy for periampullary neoplasms, involving pancreas head adenocarcinoma, malignant ampulloma and intra papillary and mucinous neoplasm
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Postoperative infectious complications at postoperative day 90 | Postoperative time until day 90
  Patients with postoperative infectious complications and compare bacteriological results of samples with bile samples.

SECONDARY OUTCOMES:
Mortality before ICU discharge | 90 days
  Mortality rate before ICU discharge
Mortality post operative day 28 | 28 days
  Mortality rate at post operative day 28
Mortality post operative day 90 | 90 days
  Mortality rate at post operative day 90

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre Pertek, MD, Study Director — CHRU Nancy
Locations (1):
- CHRU Nancy, Nancy, Grand Est, France